CLINICAL TRIAL: NCT05012423
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose, First-Time-In-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ecc0509 in Healthy Volunteers
Brief Title: FTIH Study of ECC0509 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eccogene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EC0001
Record Dates: First submitted 2021-07-22; First posted 2021-08-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Nonalcoholic Steatohepatitis; Osteoarthritis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SAD Cohorts 1 to 6: Participants Receiving Placebo (Placebo Comparator): Participants in each SAD cohort will be randomized to receive placebo.
  Interventions: Drug: Placebo
- SAD Cohorts 1 to 6: Participants receiving ECC0509 (Experimental): Participants in each SAD cohort will be randomized to receive 1 of 6 escalating doses (1 mg, 4 mg, 10 mg, 20 mg, 40 mg, or 60 mg).
  Interventions: Drug: ECC0509
- MAD Cohorts 1 to 4: Participants receiving Placebo (Placebo Comparator): Participants will be randomized to receive a once-daily dose of placebo for 14 days.
  Interventions: Drug: Placebo
- MAD Cohorts 1 to 4: Participants receiving ECC0509 (Experimental): Participants will be randomized to receive a once-daily dose of 1 of 4 escalating doses (3 mg, 10 mg, 30 mg, 60 mg) for 14 days.
  Interventions: Drug: ECC0509

INTERVENTIONS:
Drug: Placebo — Matching Placebo will be administered as oral capsules.
  Arms: SAD Cohorts 1 to 6: Participants Receiving Placebo
Drug: ECC0509 — ECC0509 1 mg and 10 mg capsules. ECC0509 will be administered as oral capsules.
  Arms: SAD Cohorts 1 to 6: Participants receiving ECC0509
Drug: Placebo — Matching Placebo will be given orally during each dosing day.
  Arms: MAD Cohorts 1 to 4: Participants receiving Placebo
Drug: ECC0509 — ECC0509 1 mg and 10 mg capsules
  Arms: MAD Cohorts 1 to 4: Participants receiving ECC0509

SUMMARY:
A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single And Multiple Ascending Dose, First-Time-In-Human Study to Assess The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ECC0509 in Healthy Volunteers.

DETAILED DESCRIPTION:
This study will be conducted in up to seven cohorts of Single Ascending Dose (SAD) & 3 cohorts of Multiple Ascending Dose (MAD). SAD will consist of a staggered dosing approach with a dose range from 1mg to 80mg. Staggered dosing approach will not be deployed for MAD cohorts with a dose range of 8mg to 40mg. In the MAD cohort, the effect of food will also be assessed by comparing the PK profile of Day 10 fed conditions against Day 14 fasted conditions.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or non-childbearing potential female
2. Age ≥18 and ≤65 years old
3. BMI ≥18.0 and ≤32.0 kg/m2
4. Male participants agree to use contraception
5. No clinically significant abnormal findings in physical examination, 12-lead electrocardiogram (ECG), laboratory tests, or medical history
6. Able to understand and sign informed consent

Key Exclusion Criteria:

1. Significant allergic reactions to any drug.
2. History of significant drug abuse or alcohol abuse within 1 year prior to screening
3. Concomitant participation in any investigational study of any nature
4. Use of any concomitant medication except for the occasional use of acetaminophen (up to 2 g daily)
5. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
6. Any clinically significant abnormal findings in the participant's physical examination, laboratory tests, pregnancy test, urine drug screen, alcohol breath test, or medical history which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, with abnormal laboratory test results, abnormal ECGs, abnormal vital signs, and abnormal physical examinations | SAD: Up to Day 8. MAD: Up to Day 21.
  Safety Assessment evaluated through adverse events, laboratory evaluations, vital signs, ECGs, and physical examination.

SECONDARY OUTCOMES:
ECC0509 PK parameters: Cl/F | SAD: Up to Day 8.
  Apparent clearance
ECC0509 PK parameters: Vz/F | SAD: Up to Day 8.
  Apparent volume of distribution
ECC0509 PK parameter: AUC0-24 | MAD: Up to Day 21
  Area under the concentration-time curve from time zero to time 24 hours
ECC0509 PK parameter: Cmax ss | MAD: Up to Day 21
  Maximal observed concentration at steady-state
ECC0509 PK parameter: Tmax ss | MAD: Up to Day 21
  Time when the maximal concentration is observed at steady-state
ECC0509 PK parameter: Tlag ss | MAD: Up to Day 21
  Time prior to the first measurable (non-zero) concentration at steady-state
ECC0509 PK parameters: Cmax | SAD: Up to Day 8. MAD: Up to Day 21
  Maximal observed concentration
ECC0509 PK parameter: Tmax | SAD: Up to Day 8. MAD: Up to Day 21
  Time when the maximal concentration is observed
ECC0509 PK parameter: AUC0-t | SAD: Up to Day 8. MAD: Up to Day 21
  Area under the curve up to the last quantifiable time-point
ECC0509 PK parameter: Cmin ss | MAD: Up to Day 21
  Minimal observed concentration at steady-state
ECC0509 PK parameter: T½ el | SAD: Up to Day 8. MAD: Up to Day 21
  Terminal elimination half-life
ECC0509 PK parameter: Kel | SAD: Up to Day 8. MAD: Up to Day 21
  Terminal elimination rate constant
ECC0509 PK parameter: Clss/F | MAD: Up to Day 21
  Apparent body clearance at steady-state
ECC0509 PK parameter: Vz ss/F | MAD: Up to Day 21
  Apparent volume of distribution at steady-state
ECC0509 PK parameter: AUC0-τ | MAD: Up to Day 21
  Area under the concentration-time curve for one dosing interval (τ) at steady state.
ECC0509 PK parameters: AUC0-inf | SAD: Up to Day 8. MAD: Up to Day 21
  Area under the concentration-time curve from time zero to infinity
ECC0509 PK parameters: Residual area | SAD: Up to Day 8. MAD: Up to Day 21
  Percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity
PD Parameter: SSAO | SAD: Up to Day 8. MAD: Up to Day 21.
  plasma semicarbazide-sensitive amine oxidase (SSAO) activity.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No